CLINICAL TRIAL: NCT06493630
Title: The Effect of Hypnobreastfeeding Education Given to Primiparas on Breastfeeding Myths, Expectations and Self-Efficacy
Brief Title: The Effect of Hypnobreastfeeding Education Given to Primiparas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Uni_emine.akca
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding; Self Efficacy; Expectations
Keywords: Primiparous pregnant women; Breastfeeding Myths
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Hypnobreastfeeding Education
  Interventions: Behavioral: Hypnobreastfeeding Education
- Control group (No Intervention): Control

INTERVENTIONS:
Behavioral: Hypnobreastfeeding Education — Hypnobreastfeeding Education: Monitoring breastfeeding myths, breastfeeding expectations and breastfeeding self-efficacy with hypnobreastfeeding education
  Arms: Experimental group

SUMMARY:
Hypnobreastfeeding is one of the education-based interventions used in this field. This study aims to evaluate the effect of hypnobreastfeeding education given to primiparous pregnant women on breastfeeding myths, breastfeeding expectations and breastfeeding self-efficacy. According to the results of the power analysis, at least 104 pregnant women, 52 experimental and 52 control, should be included in the study. Data were collected with the "Pregnant Introduction Form", "Breastfeeding Myths Scale", "Breastfeeding Expectations Scale-A" and "Prenatal Breastfeeding Self-Efficacy Scale". In the research, hypnobreastfeeding training was applied by the researcher to the primiparous pregnant women in the experimental group. The study was completed with 110 primiparous pregnant women, 54 in the experimental group and 56 in the control group.

DETAILED DESCRIPTION:
Primiparous pregnant women may need support regarding the breastfeeding process because they have not had breastfeeding experience before. Negative breastfeeding stories and misinformation can affect beliefs, attitudes, and fears about breastfeeding. Education-based interventions provided by health professionals can be beneficial in reducing false beliefs and myths about breastfeeding, reducing breastfeeding-related fears/anxious expectations, and increasing breastfeeding self-efficacy. Hypnobreastfeeding is one of the education-based interventions used in this field. This study aims to evaluate the effect of hypnobreastfeeding education given to primiparous pregnant women on breastfeeding myths, breastfeeding expectations and breastfeeding self-efficacy. According to the results of the power analysis, at least 104 pregnant women, 52 experimental and 52 control, should be included in the study. Data were collected with the "Pregnant Introduction Form", "Breastfeeding Myths Scale", "Breastfeeding Expectations Scale-A" and "Prenatal Breastfeeding Self-Efficacy Scale". In the research, hypnobreastfeeding training was applied by the researcher to the primiparous pregnant women in the experimental group. The study was completed with 110 primiparous pregnant women, 54 in the experimental group and 56 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women,
* Singleton pregnancy,
* Those with 28-32 weeks of pregnancy,
* Those who can read and write Turkish,
* Those who volunteered to participate in the study

Exclusion Criteria:

* Those with communication disabilities,
* Those with psychiatric and mental illnesses,
* Those who have an obstacle to breastfeeding,
* Those diagnosed with risky pregnancy,
* Those who have previously attended a birth preparation class,
* Those who receive breastfeeding-related training and consultancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Primiparous pregnant women
Enrollment: 110 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Myths Scale | At the end of the 1 months
  The minimum score that can be obtained from the scale is "30", the maximum score is "150", and as the score obtained from the scale decreases, breastfeeding myths levels also decrease.
Breastfeeding Expectations Scale-A | At the end of the 1 months
  The minimum score that can be obtained from the scale is "12", the maximum score is "60". Lower scores from the scale indicate more positive expectations regarding the breastfeeding experience.
Prenatal Breastfeeding Self-Efficacy Scale | At the end of the 1 months
  The minimum score that can be obtained from the scale is "20", the maximum score is "100", and as the score obtained from the scale increases, breastfeeding self-efficacy levels also increase.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, Principal Investigator — Amasya University
Locations (1):
- Emine İBİCİ AKÇA, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No